CLINICAL TRIAL: NCT06277661
Title: The Mom and Infant Outcomes (MOMI) Study: A Trial of Perinatal Outpatient Delivery Systems
Brief Title: The Mom and Infant Outcomes (MOMI) Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Shannon Gillespie, Assistant Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023H0305
Record Dates: First submitted 2024-02-07; First posted 2024-02-26 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Postpartum Depression; Postpartum Anxiety; Cardiometabolic Syndrome
Keywords: Postpartum; Mental Health; Cardiometabolic Health; Maternal-Infant Health
MeSH Terms: conditions — Depression, Postpartum; Metabolic Syndrome; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): MOMI PODS is an innovative, dyadic model of PP primary care. Informed by the Chronic Care Model (CCM) and extensive stakeholder engagement, the MOMI PODS suite of services addresses four primary domains, with a focus on preventing PRM and eliminating SES, racial, and ethnic disparities in PRM. First, MOMI PODS is a dyadic model of care, with mothers and infants cared for in tandem throughout the PP year, and beyond. Second, MOMI PODS was strategically designed to facilitate a coordinated obstetric to PP primary care transition. Third, MOMI PODS is delivered in a way that promotes tailored, evidence-based care informed by the obstetric history. Fourth, MOMI PODS systematically integrates clinical and supportive care to concurrently address clinical and psychosocial needs, with MOMI PODS engagement extending beyond the typical referral process to facilitate direct access to needed resources and empower patients.
  Interventions: Behavioral: MOMI PODS
- Enhanced Usual Care (EUC) (Active Comparator): Usual care will be enhanced in by implementing an enhanced PP care handoff as an adaptation of typical institutional discharge procedures. Specifically, under current processes, birthing parents are asked to provide the name of their infant's pediatrician during the L&D admission, must provide the name of their infant's pediatrician prior to discharge, and are assisted with identifying a pediatrician throughout this process as needed. Alternatively, under current processes, mothers are reminded to seek PP care but not required to identify the location of care or assisted with doing so. As a component of EUC, we'll provide participants with information about our 7 EUC sites and actively assist with identifying their preferred location of care and scheduling PP care. Our research team will also engage with EUC recipients throughout the study period to encourage engagement and study retention through small care packages and hand-written notes, as well as data collection.
  Interventions: Behavioral: Enhanced Usual Care (EUC)

INTERVENTIONS:
Behavioral: MOMI PODS — MOMI PODS is an innovative, dyadic model of PP primary care. Informed by the Chronic Care Model (CCM) and extensive stakeholder engagement, the MOMI PODS suite of services addresses four primary domains, with a focus on preventing PRM and eliminating SES, racial, and ethnic disparities in PRM. First, MOMI PODS is a dyadic model of care, with mothers and infants cared for in tandem throughout the PP year, and beyond. Second, MOMI PODS was strategically designed to facilitate a coordinated obstetric to PP primary care transition. Third, MOMI PODS is delivered in a way that promotes tailored, evidence-based care informed by the obstetric history. Fourth, MOMI PODS systematically integrates clinical and supportive care to concurrently address clinical and psychosocial needs, with MOMI PODS engagement extending beyond the typical referral process to facilitate direct access to needed resources and empower patients.
  Arms: Intervention
Behavioral: Enhanced Usual Care (EUC) — Usual care will be enhanced in by implementing an enhanced PP care handoff as an adaptation of typical institutional discharge procedures. Specifically, under current processes, birthing parents are asked to provide the name of their infant's pediatrician during the L&D admission, must provide the name of their infant's pediatrician prior to discharge, and are assisted with identifying a pediatrician throughout this process as needed. Alternatively, under current processes, mothers are reminded to seek PP care but not required to identify the location of care or assisted with doing so. As a component of EUC, we'll provide participants with information about our 7 EUC sites and actively assist with identifying their preferred location of care and scheduling PP care. Our research team will also engage with EUC recipients throughout the study period to encourage engagement and study retention through small care packages and hand-written notes, as well as data collection.
  Arms: Enhanced Usual Care (EUC)

SUMMARY:
The investigator's long-term goal is to mitigate pregnancy-related mortality (PRM) risk by systematically delivering integrated clinical and supportive care that is effective, equitable, and scalable. The investigator's central hypothesis is that the Multi-modal Maternal Infant Perinatal Outpatient Delivery System (MOMI PODS) will mitigate postpartum (PP) risk and reduce disparities in PP risk by improving biopsychosocial profiles and facilitating access to evidence-based clinical and supportive care. To test this hypothesis, the investigators will conduct a hybrid type 1 randomized controlled trial (RCT) of MOMI PODS versus enhanced usual care (EUC, which we will term MOMI CARE) among a total sample of 384 mother-infant dyads (192/group) following pregnancy affected by a cardiometabolic and/or mental health condition. The investigators will enroll participants on PP day 1 and collect data at baseline and 6 months and 1 year PP. The investigators will collect implementation and service data across sites.

DETAILED DESCRIPTION:
Using this data, the investigators will address the following Specific Aims:

Specific Aim 1: To evaluate the effectiveness of MOMI PODS versus EUC in mitigating cardiometabolic and mental health risk across the PP year. Hypotheses: MOMI PODS (vs. EUC) recipients will show better cardiometabolic and mental health (Primary Outcomes: higher Life's Essential 8 scores, fewer depressive and anxiety symptoms, Secondary Outcomes: fewer emergency visits and hospital readmissions).

Specific Aim 2: To identify the biopsychosocial mechanisms through which MOMI PODS affects PP cardiometabolic and mental health at the individual patient level. Hypotheses: MOMI PODS (vs. EUC) recipients will report better patient-provider relationships and less psychosocial stress and show better stress-responsive endocrine and immune profiles, which will be critical drivers of cardiometabolic and mental health.

Specific Aim 3: To determine if MOMI PODS reduces socioeconomic (SES), racial, and ethnic disparities in evidence-based PP care delivery and identify strategies to improve implementation and service outcomes. Hypotheses: MOMI PODS (vs. EUC) recipients will receive clinical and supportive care that is more adherent to evidence-based guidelines, which will reduce SES, racial, and ethnic disparities in evidence-based care. Objective: Identify strategies to improve implementation and service outcomes by evaluating fidelity, timeliness, and equity of clinical and supportive care across MOMI PODS sites.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the MOMI PODS RCT, individuals will be required to be pregnant, with a current diagnosis or history of one or more of the following reflected in the medical record or by self-report - chronic hypertension (with or without super-imposed preeclampsia); gestational hypertension; preeclampsia; eclampsia; hemolysis, elevated liver enzymes and low platelets (HELLP) syndrome; type 1 diabetes mellitus; type 2 diabetes mellitus; gestational diabetes mellitus (GDM); a depressive disorder (e.g., major depressive disorder, persistent depressive disorder) or anxiety disorder (e.g., generalized anxiety disorder, panic disorder).43-48 Inclusion criteria will also include a singleton pregnancy and medical record documentation or self-report of private or government-sponsored health insurance at the time of enrollment.

Exclusion Criteria:

Exclusion criteria will include the presence of a pre-existing, community driven MOMI PODS referral and enrollment into the program, maternal history of a seizure disorder, medical record documentation or self-report of a major complication of the infant that would be expected to preclude them from receiving or significantly delay their ability to receive outpatient pediatric care during the first year of life. Examples include but are not limited to anencephaly, myelomeningocele, esophageal atresia, gastroschisis, hypoplastic left heart syndrome, transposition of the great arteries, or tetralogy of Fallot. Exclusion criteria will also include the presence of a major genetic disorder among the infant that would be expected to preclude them from receiving or significantly delay their ability to receive outpatient pediatric care during the first year of life. Examples include but are not limited to trisomy 13, or trisomy 18 (trisomy 21 is not an exclusion criteria).

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 384 (Estimated)
Dates: Start 2024-06-27 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in Life's Essential 8 (LE8) Composite Score | Baseline (T1) to 6 months postpartum (T2)
  Higher scores=better health (0-100). 0-100 points for each domain. Total divided by 8. Diet (Mediterranean Eating Pattern for Americans score): 100=15-16; 80=12-14; 50=8-11; 25=4-7; 0=0-3; Physical Activity (min. moderate+/week): 100=>=150; 90=120-149; 80=90-119; 60=60-89; 40=30-59; 20=1-29; 0=0; Nicotine: 100=Never; 75=Former, quit >=5y; 50=Former, quit 1-<5y; 25=Former, quit <1y or vaping; 0=Current; -20 living with indoor smoker; Sleep (avg. hrs./night): 100=7<9; 90=9-<10; 70=6-<7; 40=5-<6 or >=10; 20=4-<5; 0=<4; body mass index (kg/m2): 100=<25; 70=25-29.9; 30=30-34.9; 15=35-39.9; 0=>=40; Non-HDL mg/dL: 100=<130; 60=130-159; 40=160-189; 20=190-219; 0=>=220; -20 if treated; Glucose (Diabetes/HbA1c): 100=No/<5.7; 60=No/5.7-6.4; 40=Yes/<7; 30=Yes/7-7.9; 20=Yes/8-8.9; 10=Yes/9-9.9; 0=Yes/>=10; Blood pressure: 100=<120/<80; 75=120-129/<80; 50=130-139 or 80-89; 25=140-159 or 90-99; 0=>=160 or >=100; -20 if treated
Change in Life's Essential 8 (LE8) Composite Score | 6 months postpartum (T2) to 12 months postpartum (T3)
  Higher scores=better health (0-100). 0-100 points for each domain. Total divided by 8. Diet (Mediterranean Eating Pattern for Americans score): 100=15-16; 80=12-14; 50=8-11; 25=4-7; 0=0-3; Physical Activity (min. moderate+/week): 100=>=150; 90=120-149; 80=90-119; 60=60-89; 40=30-59; 20=1-29; 0=0; Nicotine: 100=Never; 75=Former, quit >=5y; 50=Former, quit 1-<5y; 25=Former, quit <1y or vaping; 0=Current; -20 living with indoor smoker; Sleep (avg. hrs./night): 100=7<9; 90=9-<10; 70=6-<7; 40=5-<6 or >=10; 20=4-<5; 0=<4; body mass index (kg/m2): 100=<25; 70=25-29.9; 30=30-34.9; 15=35-39.9; 0=>=40; Non-HDL mg/dL: 100=<130; 60=130-159; 40=160-189; 20=190-219; 0=>=220; -20 if treated; Glucose (Diabetes/HbA1c): 100=No/<5.7; 60=No/5.7-6.4; 40=Yes/<7; 30=Yes/7-7.9; 20=Yes/8-8.9; 10=Yes/9-9.9; 0=Yes/>=10; Blood pressure: 100=<120/<80; 75=120-129/<80; 50=130-139 or 80-89; 25=140-159 or 90-99; 0=>=160 or >=100; -20 if treated
Change in Life's Essential 8 (LE8) Composite Score | Baseline (T1) to 12 months postpartum (T3)
  Higher scores=better health (0-100). 0-100 points for each domain. Total divided by 8. Diet (Mediterranean Eating Pattern for Americans score): 100=15-16; 80=12-14; 50=8-11; 25=4-7; 0=0-3; Physical Activity (min. moderate+/week): 100=>=150; 90=120-149; 80=90-119; 60=60-89; 40=30-59; 20=1-29; 0=0; Nicotine: 100=Never; 75=Former, quit >=5y; 50=Former, quit 1-<5y; 25=Former, quit <1y or vaping; 0=Current; -20 living with indoor smoker; Sleep (avg. hrs./night): 100=7<9; 90=9-<10; 70=6-<7; 40=5-<6 or >=10; 20=4-<5; 0=<4; body mass index (kg/m2): 100=<25; 70=25-29.9; 30=30-34.9; 15=35-39.9; 0=>=40; Non-HDL mg/dL: 100=<130; 60=130-159; 40=160-189; 20=190-219; 0=>=220; -20 if treated; Glucose (Diabetes/HbA1c): 100=No/<5.7; 60=No/5.7-6.4; 40=Yes/<7; 30=Yes/7-7.9; 20=Yes/8-8.9; 10=Yes/9-9.9; 0=Yes/>=10; Blood pressure: 100=<120/<80; 75=120-129/<80; 50=130-139 or 80-89; 25=140-159 or 90-99; 0=>=160 or >=100; -20 if treated
Change in Patient Health Questionnaire-9 (PHQ-9) Score | Baseline (T1) to 6 months postpartum (T2)
  We will assess mental health by self-report using the Patient Health Questionnaire-9 (PHQ-9), with higher scores indicative of more depressive symptoms (range 0-27).
Change in Patient Health Questionnaire-9 (PHQ-9) Score | 6 months postpartum (T2) to 12 months postpartum (T3)
  We will assess mental health by self-report using the Patient Health Questionnaire-9 (PHQ-9), with higher scores indicative of more depressive symptoms (range 0-27).
Change in Patient Health Questionnaire-9 (PHQ-9) Score | Baseline (T1) to 12 months postpartum (T3)
  We will assess mental health by self-report using the Patient Health Questionnaire-9 (PHQ-9), with higher scores indicative of more depressive symptoms (range 0-27).
Change in Generalized Anxiety Disorder-7 (GAD-7) Score | Baseline (T1) to 6 months postpartum (T2)
  We will assess mental health by self-report using the Generalized Anxiety Disorder-7 (GAD-7), with higher scores indicative of more anxiety symptoms (range 0-21).
Change in Generalized Anxiety Disorder-7 (GAD-7) Score | 6 months postpartum (T2) to 12 months postpartum (T3)
  We will assess mental health by self-report using the Generalized Anxiety Disorder-7 (GAD-7), with higher scores indicative of more anxiety symptoms (range 0-21).
Change in Generalized Anxiety Disorder-7 (GAD-7) Score | Baseline (T1) to 12 months postpartum (T3)
  We will assess mental health by self-report using the Generalized Anxiety Disorder-7 (GAD-7), with higher scores indicative of more anxiety symptoms (range 0-21).

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with the NIH Policy for Data Management and Sharing, we've carefully considered the data expected to be generated and the best approach to maximize the appropriate sharing of scientific data while also protecting the privacy of human subjects participating in research. We expect remnant biospecimens to be minimal after study execution and will therefore not submit biospecimens. Also of note, obstetric complications, postnatal complications, severe maternal morbidity (SMM), and pregnancy-related mortality (PRM) are rare occurrences. Details surrounding this information are publicly available in birth and death certificates and could be aligned with other information to identify a research participant. Thus, to protect participant privacy, we do not plan to share raw data but will produce collapsed variables for data sharing.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be made available at the time of associated publications, or the end of the performance period, whichever comes first. Data and Specimen Hub (DASH) considers submitted datasets to be permanently available.
Access Criteria: All requests for data through DASH is routed through the National Institute of Child Health and Human Development (NICHD) DASH Data and Biospecimen Access Committee. This committee reviews these requests and determines whether the proposed use is scientifically and ethically appropriate and does not conflict with data use limitations identified by the submitting institution. If deemed necessary, the committee will obtain additional approvals from the study-specific entity, such as the Multiple Principle Investigators (MPIs).